CLINICAL TRIAL: NCT04067154
Title: Does a Bedside Method for Describing Functional Gas Exchange Compare Well With Anatomical Description Via CT Scans, and Could it Predict the Effects of Recruitment and Ventilation/Perfusion Mismatch Improvement
Brief Title: Gas Exchange and CT Effects of PEEP in ARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Mauro Panigada, Does a bedside method for describing functional gas exchange compare well with anatomical description via CT scans, and could it predict the effects of recruitment and ventilation/perfusion mismatch improvement., Policlinico Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2425
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: ARDS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ALPE-TAC (Experimental): ARDS patients on mechanical ventilation. Measurement of CT scan at PEEP of 5, 20 and 45 cm H2O to evaluate potential for recruitment and measurement of gas exchange by model-based method and FiO2 titration at PEEP of 5 and 20 cm H2O
  Interventions: Diagnostic Test: ALPE

INTERVENTIONS:
Diagnostic Test: ALPE — Measurement of CT scan at PEEP of 5, 20 and 45 cm H2O Measurement of gas exchange by model-based method and FiO2 titration at PEEP of 5 and 20 cm H2O

SUMMARY:
The study aims to investigate the association between effects of PEEP on gas exchange model parameters and CT scan results

DETAILED DESCRIPTION:
In ARDS patients on mechanical ventilation, we will compare model-based estimation of gas exchange parameters (shunt, ventilation/perfusion mismatch) with CT-based estimation of effects of low and high PEEP

ELIGIBILITY:
Inclusion Criteria:

- ARDS patients requiring mechanical ventilation

Exclusion Criteria:

* <18 years old
* Requirement of extracorporal life support
* Hemodynamic instability
* Barotrauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2014-08-01 (Actual); Study Completion 2014-08-01 (Actual)

PRIMARY OUTCOMES:
Gas Exchange and lung recruitability at diferent PEEP levels | Approximately two hours
  Gas exchange (At PEEP 5 and 20 cm H2O), CT scan (At PEEP 5, 20 and 45 cm H2O)

SECONDARY OUTCOMES:
Physiologic Parameter 1 | Approximately two hours
  Hemodynamic assessment at different PEEP levels
Physiologic Parameter 2 | Approximately two hours
  Respiratory mechanics at different PEEP levels

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, MI, Italy

REFERENCES:
- [Derived] Karbing DS, Panigada M, Bottino N, Spinelli E, Protti A, Rees SE, Gattinoni L. Changes in shunt, ventilation/perfusion mismatch, and lung aeration with PEEP in patients with ARDS: a prospective single-arm interventional study. Crit Care. 2020 Mar 23;24(1):111. doi: 10.1186/s13054-020-2834-6. PMID 32293506